CLINICAL TRIAL: NCT04395248
Title: An Investigation of Optimal Anesthesia for Morbidly Obese Patients Undergoing Bariatric Surgery: A Randomized Controlled Trial
Brief Title: Optimal Anesthesia for Morbidly Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, YingHsuanTai, Principal Investigator, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: N202002076
Record Dates: First submitted 2020-05-11; First posted 2020-05-20 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Obesity; Anesthesia
Keywords: Obesity; Anesthesia; Enhanced recovery after surgery; Difficult intubation; Preoxygenation; Depth of anesthesia; High-flow nasal cannula
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Risk factors of difficult intubation (Active Comparator): Appearance anpalpationpalpationpalpationd ultrasound features for predicting difficult laryngoscopy intubation
  Interventions: Procedure: Exploring potential risk factors of difficult intubation using ultrasound
- Radial artery cannulation using ultrasound or blind palpation (Active Comparator): In the ultrasound group, a linear vascular probe in the frequencies 5 to 13 MHz (GE 12L-RS, GE Healthcare, Chicago, IL, USA) of portable ultrasound device (LOGIQTM, GE Healthcare, Chicago, IL, USA) will be applied to the skin to localize the radial artery and a 20-gauge catheter will be inserted distal to the transducer and directed according to the ultrasound image.
  Interventions: Procedure: Radial artery catheterization using ultrasound guidance or blind palpation
- Preoxygenation using high-flow nasal cannula or facemask (Active Comparator): In the HFNC group, preoxygenation will be performed using HFNC (Optiflow™, Fisher & Paykel Healthcare, Auckland, NZ), nasal prongs set at 30 L/min flow of heated and humidified 100% oxygen. In the facemask group, patients will breath spontaneously with an anesthetic facemask and 100% oxygen 15 L/min. Gas flow for HFNC or facemask can be adjusted depending on patients' tolerance. During laryngoscopy intubation, HFNC will be left in place with the nasal flow escalated to 50 L/min of 100% oxygen in order to achieve apneic oxygenation. In the facemask group, the facemask will be removed when apnea occurs.
  Interventions: Device: Comparing the effectiveness of preoxygenation between high-flow nasal cannula and facemask
- Type of volatile anesthetics and M-Entropy guidance (Active Comparator): Patients will be randomized by a computer-generated list into one of the four groups, desflurane with usual care (N=20), desflurane with M-Entropy guidance (N=20), sevoflurane with usual care (N=20), and sevoflurane with M-Entropy guidance (N=20).
  Interventions: Drug: Type of volatile anesthetics and M-Entropy guidance of anesthesia depth

INTERVENTIONS:
Procedure: Exploring potential risk factors of difficult intubation using ultrasound — Before surgery, ultrasound will be used to assess pretracheal soft tissue depth and height and width of tongue base. The distance from the skin to the anterior aspect of the trachea will be measured at three levels: vocal cords, thyroid isthmus, and suprasternal notch. With the patient in a seated position, the convex transducer of a portable ultrasound device (LOGIQTM, GE Healthcare, Chicago, IL, USA) will be introduced to the skin of the neck in the submental region coronally, immediately cephalad to the body of the hyoid bone, and then in the area between the hyoid bone and the symphysis of the mandible. Maximal width of tongue base, tongue base height, and maximal height of mid-tongue will be measured. The laryngoscopy intubation will be performed using a size-3 or -4 Macintosh (Rüsch Inc., Duluth, GA, USA) blade and a styletted endotracheal tube. The laryngoscopic view will be graded according to Cormack and Lehane's classification with external laryngeal pressure applied.
  Arms: Risk factors of difficult intubation
Procedure: Radial artery catheterization using ultrasound guidance or blind palpation — For all patients, the wrist will be extended and taped to a board to maintain wrist extension. All patients will receive local skin anesthesia at the anticipated puncture site. All radial artery catheterizations will be performed by anesthesiology residents with similar levels of experience in both blind-palpation and ultrasound-guided radial arterial catheterization. In the ultrasound group, a linear vascular probe of portable ultrasound device (LOGIQTM, GE Healthcare, Chicago, IL, USA) will be applied to the skin to localize the radial artery and a 20-gauge catheter will be inserted distal to the transducer and directed according to the ultrasound image. In the palpation group, the radial artery will be identified by palpation, and the cannula will be directed by continuous or intermittent palpation of arterial pulsation. An attempt is defined as a new penetration of the skin with the needle, followed by an unlimited number of subcutaneous needle redirections.
  Arms: Radial artery cannulation using ultrasound or blind palpation
Device: Comparing the effectiveness of preoxygenation between high-flow nasal cannula and facemask — In the HFNC group, preoxygenation will be performed using HFNC (Optiflow™, Fisher & Paykel Healthcare, Auckland, NZ), nasal prongs set at 30 L/min flow of heated and humidified 100% oxygen. In the facemask group, patients will breath spontaneously with an anesthetic facemask and 100% oxygen 15 L/min. Gas flow for HFNC or facemask can be adjusted depending on patients' tolerance. During laryngoscopy intubation, HFNC will be left in place with the nasal flow escalated to 50 L/min of 100% oxygen in order to achieve apneic oxygenation. In the facemask group, the facemask will be removed when apnea occurs. After tracheal intubation, correct placement of the endotracheal tube will be confirmed by capnography and the nasal prongs of the HFNC group will be removed.
  Arms: Preoxygenation using high-flow nasal cannula or facemask
Drug: Type of volatile anesthetics and M-Entropy guidance of anesthesia depth — At the operating room, a M-Entropy™ sensor and S/5™ module (GE Healthcare, Helsinki, Finland) will be applied to all patients' forehead before induction of anesthesia according to the manufacturer's recommendations. Patients will be randomized to Sevoflurane or Desflurane as the single volatile anesthetics for general anesthesia.
  Besides, patients will be randomized to M-Entropy group or controls. In the M-Entropy group, dosage of volatile anesthetics will be adjusted to achieve the Response and State Entropy value between 40 and 60 from the start of anesthesia to the end of surgery. In the usual care group, dosage of volatile anesthetics will be titrated according to clinical judgment. M-Entropy monitoring will be continued in the usual care group, but the Entropy number and EEG waveform will be concealed from the anesthetist in charge.
  Arms: Type of volatile anesthetics and M-Entropy guidance

SUMMARY:
Obese patients have a higher risk of anesthesia compared to the non-obese, including difficult intubation, rapid desaturation, difficult vascular access, and delayed recovery from anesthesia. This study aims to investigate the optimal anesthesia strategy for morbidly obese patients undergoing bariatric surgery in airway management, preoxygenation, arterial cannulation, and type of volatile anesthetic with M-Entropy guidance. The investigators will conduct a two-year clinical trial using permuted block randomization to evaluate multiple outcomes in patients undergoing laparoscopic sleeve gastrectomy (LSG) at Shuang Ho Hospital, Taipei Medical University. Particularly, the investigators will explore the role of ultrasound, an easily accessible modality for anesthesiologists, in examining upper airway anatomy and guiding arterial cannulation. The investigators will also assess the effectiveness of high-flow nasal cannula as a preoxygenation tool in preventing desaturation.

DETAILED DESCRIPTION:
The investigators will conduct a clinical trial using permuted block randomization and conforming to the CONSORT Statement to investigate multiple clinical outcomes in obese patients undergoing LSG at Shuang Ho Hospital, Taipei Medical University, New Taipei City, Taiwan. Three randomizations will be conducted, including radial artery catheterization using ultrasound guidance or blind palpitation, preoxygenation using HFNC or CPAP, and volatile anesthesia with desflurane or sevoflurane with or without M-Entropy guidance. A computer-generated list of randomizations (Research Randomizer, www.randomizer.org) will be used for these group allocations.

1. Exploring potential risk factors of difficult intubation using ultrasound: A prospective single-blind cohort study

   Before surgery, all enrolled patients will be examined for appearance features regarding difficult airway, including interincisor distance (< 3 cm or not), mentohyoid distance, thyromental distance (< 6.5 cm or not), neck movement (< 80 degrees or not), neck circumference measured at the thyroid cartilage (> 43 cm or not), modified Mallampati score, upper lip bite test, and mandibular prognathism test. Besides, ultrasound will be used to assess upper airway anatomy, including pretracheal soft tissue depth27 and height and width of tongue base. Regarding pretracheal soft tissue depth, the distance from the skin to the anterior aspect of the trachea will be measured at three levels: vocal cords, thyroid isthmus, and suprasternal notch. The amount of soft tissue at each zone is calculated by averaging the amounts of soft tissue in millimeters obtained in the central axis of the neck and 15 millimeters to the left and right of the central axis.

   Moreover, the increased tongue volume and deposition of fat at the base of tongue in obese people has been shown to be highly associated with risk of obstructive sleep apnea. To measure the anatomy of tongue base, with the patient in a seated position, the convex transducer in the frequencies 1.5 to 5.0 MHz (GE C1-5-RS, GE Healthcare, Chicago, IL, USA) of a portable ultrasound device (LOGIQTM, GE Healthcare, Chicago, IL, USA) will be introduced to the skin of the neck in the submental region coronally, immediately cephalad to the body of the hyoid bone, and then in the area between the hyoid bone and the symphysis of the mandible. The patients will be instructed to avoid tongue movements, swallowing, or talking. Maximal width of tongue base, tongue base height, and maximal height of mid-tongue will be measured. The same anesthesiologist will perform all ultrasound measurements before surgery. Upon arrival at operating room, patients will be initially placed in a ramped position and then moved into a reverse Trendelenburg position to achieve a 30-degree incline of the thorax before preoxygenation.

   After induction of anesthesia, another anesthesiologist, blinded to all preoperative evaluation, will perform all laryngoscopies in this study. The laryngoscopy intubation will be performed using a size-3 or -4 Macintosh (Rüsch Inc., Duluth, GA, USA) blade and a styletted endotracheal tube. The laryngoscopic view will be graded according to Cormack and Lehane's classification with external laryngeal pressure applied.59 Laryngoscopy views graded as III or IV are defined as difficult. In case of failed direct laryngoscopy despite external laryngeal manipulation in the first attempt, video-assisted laryngoscope GlideScope® (Verathon Medical, Bothell, WA, USA) will be used as an intubation rescue technique. The video-assisted laryngoscope will be kept on standby at the operating room before induction. The correct placement of the endotracheal tube will be confirmed by capnography.
2. Radial artery catheterization using ultrasound guidance or blind palpation: An open-label randomized controlled trial

   Before surgery, the investigators will use a portable ultrasound device (LOGIQTM, GE Healthcare, Chicago, IL, USA) to measure the skin-to-artery distance of common sites of arterial cannulation of all enrolled patients, including radial artery, brachial artery and dorsalis pedis artery. Patients will be randomized in a ratio of 1:1 into ultrasound group (N=40) or palpation group (N=40). Radial artery cannulation will be performed using a radial artery catheterization kit (Arrow International Inc, Reading, PA, USA). For all patients, the wrist will be extended and taped to a board to maintain wrist extension, and the skin near the puncture site will be cleaned with chlorhexidine according to standard protocol. Allen test will be used to assess the vascular patency of the hand before cannulation of the radial artery. All patients will receive local skin anesthesia at the anticipated puncture site. All radial artery catheterizations will be performed by trained year 1 or 2 anesthesiology residents with similar levels of experience in both blind-palpation and ultrasound-guided radial arterial catheterization. All residents have performed at least 5 blind-palpation and 5 ultrasound-guided radial arterial catheterizations prior to the study.

   In the ultrasound group, a linear vascular probe in the frequencies 5 to 13 MHz (GE 12L-RS, GE Healthcare, Chicago, IL, USA) of portable ultrasound device (LOGIQTM, GE Healthcare, Chicago, IL, USA) will be applied to the skin to localize the radial artery and a 20-gauge catheter will be inserted distal to the transducer and directed according to the ultrasound image. Start time is defined as the time when the ultrasound probe is placed on the wrist. In the palpation group, the radial artery will be identified by palpation, and the cannula will be directed by continuous or intermittent palpation of arterial pulsation. The attending anesthesiologist will supervise the resident and act as the second operator if needed. An attempt is defined as a new penetration of the skin with the needle, followed by an unlimited number of subcutaneous needle redirections. Clinical judgment by the supervising anesthesiologist is used to determine the time allowed for an attempt, number of attempts allowed, and changes to a new site. The start time is defined when the operator's finger is initially placed on the patient's wrist. The end point for both methods is when the arterial catheter is successful placed.
3. Comparing the effectiveness of preoxygenation between high-flow nasal cannula (HFNC) and facemask: A single-blind randomized controlled trial

   Patients will be randomized in an allocation ratio of 1:1 into HFNC group (N=40) or facemask group (N=40). Preoxygenation will be performed according to the randomization group for a 5-minute duration. In the HFNC group, preoxygenation will be performed using HFNC (Optiflow™, Fisher & Paykel Healthcare, Auckland, NZ), nasal prongs set at 30 L/min flow of heated and humidified 100% oxygen. In the facemask group, patients will breath spontaneously with an anesthetic facemask and 100% oxygen 15 L/min. Gas flow for HFNC or facemask can be adjusted depending on patients' tolerance. During laryngoscopy intubation, HFNC will be left in place with the nasal flow escalated to 50 L/min of 100% oxygen in order to achieve apneic oxygenation. In the facemask group, the facemask will be removed when apnea occurs. After tracheal intubation, correct placement of the endotracheal tube will be confirmed by capnography and the nasal prongs of the HFNC group will be removed. If desaturation (SpO2 < 92%) occurs, patients will be then administered 100% O2, and the recruitment maneuver (peak airway pressure 40 cm H2O for 10 seconds) will be applied until SpO2 restores to baseline values.
4. The effect of type of volatile anesthetics and M-Entropy guidance of anesthesia depth on postoperative recovery: A double-blind randomized controlled trial

Patients will be randomized by a computer-generated list into one of the four groups, desflurane with usual care (N=20), desflurane with M-Entropy guidance (N=20), sevoflurane with usual care (N=20), and sevoflurane with M-Entropy guidance (N=20). At the operating room, a M-Entropy™ sensor and S/5™ module (GE Healthcare, Helsinki, Finland) will be applied to all patients' forehead before induction of anesthesia according to the manufacturer's recommendations. This will be connected to a M-Entropy Monitor that will be concealed from the patients and operators.

In the M-Entropy group, dosage of volatile anesthetics will be adjusted to achieve the Response and State Entropy value between 40 and 60 from the start of anesthesia to the end of surgery. In the usual care group, dosage of volatile anesthetics will be titrated according to clinical judgment. This will be to maintain arterial pressure within 20% range of the baseline and the heart rate within the range 50 to 100 beats/min. In case of signs of inadequate anesthesia (e.g. movement, cough and swallowing), anesthetic dose will be increased. M-Entropy monitoring will be continued in the usual care group, but the Entropy number and EEG waveform will be concealed from the anesthetist in charge. Entropy values, hemodynamic, and expiratory gas data will be recorded in 5-min intervals. In all patients, cessation of general anesthesia will be timed to facilitate early awakening after wound closure. All patients will be decurarized from rocuronium-induced neuromuscular blockade with sugammadex dosed at 2 mg/kg ideal body weight + 40%.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 65 years
* BMI ≥ 30 kg/m2
* Undergoing laparoscopic sleeve gastrectomy at Shuang-Ho Hospital, Taiwan

Exclusion Criteria:

* Severe cardiopulmonary disease
* Psychiatric disorder
* History of head and neck surgery or radiation therapy
* Cervical spine injury
* Renal insufficiency (estimated creatinine clearance < 60 ml/min)
* SpO2 < 90% in room air
* Hemodynamic instability
* Preexisting arterial catheterization during the same visit within 7 days
* Patient refusal

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of difficult laryngoscopy | One day before surgery to tracheal intubation
  The laryngoscopic view will be graded according to Cormack and Lehane's classification with external laryngeal pressure applied. Grade 1: Most of the glottis is visible; Grade 2: At best almost half of the glottis is seen, at worst only the posterior tip of the arytenoids is seen; Grade 3: Only the epiglottis is visible; Grade 4: No laryngeal structures are visible.
First-attempt success rate for arterial cannulation | Before induction of anesthesia
  An attempt is defined as a new penetration of the skin with the needle, followed by an unlimited number of subcutaneous needle redirections.
PaO2 after preoxygenation | Before induction of anesthesia
  Arterial blood gas will be analyzed promptly after 5-min preoxygenation.
Time to spontaneous eye opening | The period from discontinuation of volatile anesthetics to spontaneous eye opening, an average of 15 minutes
  The interval from discontinuation of volatile anesthetics to spontaneous eye opening

SECONDARY OUTCOMES:
First-attempt success rate for intubation | After induction of anesthesia
  As title
Time to successful intubation | After induction of anesthesia
  After tracheal intubation, correct placement of the endotracheal tube will be confirmed by capnography.
Time to successful arterial catheterization | Before induction of anesthesia
  The interval from the finger or ultrasound probe touching the skin to successful arterial catheterization
Number of attempts for arterial cannulation | Before induction of anesthesia
  An attempt is defined as a new penetration of the skin with the needle, followed by an unlimited number of subcutaneous needle redirections.
Number of sites and catheters used for arterial cannulation | Before induction of anesthesia
  As title
Relevant complications of arterial cannulation | Before induction of anesthesia
  Including pain, ultrasound-measured hematoma, arterial vasospasm, and arterial occlusion.
SpO2 before and after preoxygenation | Before induction of anesthesia
  As title
Desaturation event during intubation | After induction of anesthesia
  Defined as SpO2 < 92%
The lowest SpO2 during intubation | After induction of anesthesia
  As title
PaCO2 before and after preoxygenation | Before induction of anesthesia
  Arterial blood gas will be analyzed twice before and after preoxygenation
Patient comfort levels | Before induction of anesthesia
  Measured by 10-point Likert scale, 0 minimal comfort and 10 maximal comfort
Time to tracheal extubation | The period from discontinuation of volatile anesthetics to tracheal extubation, an average of 25 minutes
  The interval from discontinuation of volatile anesthetics to tracheal extubation
Time to orientation in time and place | The period from discontinuation of volatile anesthetics to orientation in time and place, an average of 20 minutes
  The interval from discontinuation of volatile anesthetics to orientation in time and place
Time to leave operating room | The period from discontinuation of volatile anesthetics to leaving operating room, an average of 30 minutes
  The interval from discontinuation of volatile anesthetics to leaving operating room
Event of emergence agitation | During or after tracheal intubation at the end of surgery
  Measured by Richmond Agitation-Sedation Scale, classifying into combative, very agitated, agitated, restless, alter and calm, and drowsy

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Hsuan Tai, M.D., M.Sc., Principal Investigator — Department of Anesthesiolgy, Shuang-Ho Hospital, Taipei Medical University, Taiwan
Locations (1):
- Department of Anesthesiology, Shuang-Ho Hospital, Taipei Medical University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu YM, Su YH, Huang SY, Wang CW, Shen SC, Chen JT, Lo PH, Cherng YG, Wu HL, Tai YH. Morphometric and ultrasonographic determinants of difficult laryngoscopy in obese patients: A prospective observational study. J Chin Med Assoc. 2022 May 1;85(5):571-577. doi: 10.1097/JCMA.0000000000000721. Epub 2022 May 2. PMID 35385418

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT04395248/Prot_SAP_000.pdf